CLINICAL TRIAL: NCT06324526
Title: What is the Effect of Bariatric Surgery on Health-related Quality of Life? Analysis of the United Kingdom National Bariatric Surgery Registry
Brief Title: Obesity and Health-related Quality of Life in Patients Receiving Bariatric Surgery in the UK
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Collaborators: University of Oxford (Other)
Responsible Party: Sponsor
Other Study IDs: 070324QL
Record Dates: First submitted 2024-03-15; First posted 2024-03-22 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Quality of Life; Obesity, Morbid; Bariatric Surgery Candidate
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- People undergoing bariatric surgery: People under going primary bariatric surgery between 1st June 2017 and 23rd November 2022 with complete health-related quality of life records (EQ-5D) with one pre-operative and at least one follow-up record within 1 year of surgery.

SUMMARY:
United Kingdom National Bariatric Surgery Registry (NBSR) records between 1st June 2017 and 23rd November 2022 were used to identify people undergoing primary bariatric (weight-loss) surgery. People undergoing primary bariatric (weight-loss) surgery with one baseline and at least one follow-up visit within one year from surgery were included. Statistical models were used to estimate the relationship between quality of life as assessed by a questionnaire and body mass index at baseline and over time.

DETAILED DESCRIPTION:
Previous small studies investigating health-related quality of life (HRQoL) following bariatric surgery have demonstrated heterogenous effects. Estimated changes in HRQoL are used to evaluate both clinical- and cost-effectiveness of interventions; which in turn informs commissioning decisions. Understanding HRQoL of patients undergoing bariatric surgery is therefore important for both clinical practice and policymaking.

This study aimed to use National Bariatric Surgery Registry (NBSR) records to investigate the relationship between weight and HRQoL in people undergoing bariatric surgery in the UK. The NBSR is an anonymised, bespoke record of bariatric cases carried out within the National Health Service (NHS) in the UK and Ireland. The analysis plan was prospectively published in March 2022, and it is available here: https://osf.io/6t9rg/.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18 years or older)
* undergoing primary bariatric surgery
* with both baseline (pre-operative) and at least one follow-up record.

Exclusion Criteria:

* people undergoing revision surgery
* records that did not include complete EQ-5D scoring (all 5 domains).
* records with implausible values, defined as: BMI <25 kg/m2 or >100 kg/m2; height <1m or >2.5m; weight <50kg or >400kg; age>100 years.
* records greater than 12 months from surgery date

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Records were selected from the NBSR (National Bariatric Surgery Registry) which is an anonymised, bespoke record of bariatric cases carried out within the National Health Service (NHS) in the UK and Ireland.
Sampling Method: Non-Probability Sample
Enrollment: 2160 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2022-11-23 (Actual); Study Completion 2022-11-23 (Actual)

PRIMARY OUTCOMES:
EQ-5D (EuroQol Five Dimension) | up to 1 year post-operatively
  EuroQol Five Dimension 5-level (validated measure for health-related quality of life). This is a validated measure of health-related quality of life (HRQoL) (see references).
  Subjects are asked to rate the level of problems they experience related to 5 domains of HRQoL (mobility, self care, usual activities, pain/discomfort and anxiety/depression). There are 5 values to choose from in each domain (e.g. no problem, slight problem, moderate problem, severe problem, unable to). A higher score indicates a worse quality of life.
  EQ-5D scores are converted to overall utilities by averaging domains and weighting by the general public's valuation of the domains. A higher overall utility score for EQ-5D represents better HRQoL.
BMI | up to 1 year post-operatively
  Body mass index in kg/m2

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Surgery and Cancer, Imperial College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
There are restrictions on the availability of data for this study, due to the initial patient consent forms, which only allow the sharing of data for research purposes. Researchers wishing to access an anonymized dataset can apply to the corresponding author.

REFERENCES:
- [Background] Herdman M, Gudex C, Lloyd A, Janssen M, Kind P, Parkin D, Bonsel G, Badia X. Development and preliminary testing of the new five-level version of EQ-5D (EQ-5D-5L). Qual Life Res. 2011 Dec;20(10):1727-36. doi: 10.1007/s11136-011-9903-x. Epub 2011 Apr 9. PMID 21479777
- [Derived] Buckell J, Small PK, Jebb SA, Aveyard P, Khan O, McGlone ER; NBSR Collaborators. What is the effect of bariatric surgery on health-related quality of life in people with obesity? Observational cohort analysis of the United Kingdom National Bariatric Surgery Registry. Int J Surg. 2024 Nov 1;110(11):6898-6905. doi: 10.1097/JS9.0000000000002044. PMID 39172711
- See also: analysis plan — http://osf.io/6t9rg/